CLINICAL TRIAL: NCT06671639
Title: Stanford Program to Accelerate Robotic Children's Surgery
Acronym: SPARCS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 78052
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Sleeve Gastrectomy; Cholecystectomy; Splenectomy; Hysterectomy; Endometriosis; Ureteral Re-implant; Cervical and Thoracic Tracheoplasty; Thymectomy; Lobectomy/wedge Lung Resection; Lung Segmentectomy; Bronchoplasty; Endoscopic Laryngeal/Pharyngeal Suturing; Vocal Feminization; Laryngeal Cleft Repair; Endolaryngeal Adjacent Tissue Transfer; Pharyngoplasty; Ileocolonic Resections; Laryngoplasty; Proctectomy with Ileal Pouch-Anal Anastomosis
Keywords: Robotic Surgery; Pediatric Robotic Surgery
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm 1 (Experimental): Arm 1 includes procedures to be performed robotically that have an adult model or already established preclinical evidence including: Sleeve Gastrectomy, Cholecystectomy, Splenectomy, Hysterectomy, endometriosis, ureteral re-implant, and cervical and thoracic tracheoplasty, thymectomy, lobectomy/wedge lung resection, lung segmentectomy
  Interventions: Device: da Vinci Xi Robotic Surgery System
- Arm 2 (Experimental): Arm 2 will be performed after all patients in Arm 1 have completed their procedures and where additional preclinical performance testing is required, including: Bronchoplasty, Endoscopic Laryngeal/Pharyngeal Suturing, including: Vocal Feminization, Laryngeal Cleft Repair, Endolaryngeal Adjacent Tissue Transfer, Pharyngoplasty; Ileocolonic Resections; Laryngoplasty with or without Graft; Proctectomy with Ileal Pouch-Anal Anastomosis (IPAA)
  Interventions: Device: da Vinci Xi Robotic Surgery System

INTERVENTIONS:
Device: da Vinci Xi Robotic Surgery System — The da Vinci Xi Surgical System is a software-controlled, electro-mechanical system designed for surgeons to perform minimally invasive surgery. It consists of a Surgeon Console, a Patient Cart, and a Vision Cart, and is used with a Camera Instrument and EndoWrist Xi instruments and accessories.
  The surgeon seated at the surgeon console controls all movement of the EndoWrist Xi instruments and Camera Instrument using two master controls and a set of foot pedals. The surgeon views the three-dimensional endoscopic image on a high-resolution stereo viewer (3D viewer), which provides him/her/they a view of patient anatomy and instrumentation, along with icons and other user interface features. The Vision Cart includes the supporting electronic and video processing equipment for the system.

SUMMARY:
The goal of this clinical trial is to provide additional data to confirm safety and performance of the da Vinci Xi Surgical System in a human clinical setting. This pilot study is intended to provide an initial assessment to evaluate the feasibility, safety, and effectiveness for the utilization of the da Vinci Xi on pediatric and adolescent patients. This clinical trial will be conducted under the auspices of Stanford University's IRB approval.

DETAILED DESCRIPTION:
Advancements in robotic technology have facilitated the expansion of pediatric robotic surgery, enabling surgeons to perform increasingly complex procedures with greater precision and efficiency. Improved robotic platforms, enhanced imaging modalities, and innovative surgical techniques have contributed to the evolution of pediatric robotic surgery. Moreover, the development of specialized instruments and accessories tailored to pediatric patients, while in limited fashion, has further enhanced the safety and feasibility of robotic-assisted procedures in this population.

The objective of this clinical study is to provide preliminary evidence showcasing that the da Vinci Xi Surgical System is substantially equivalent to existing surgical techniques for the performance of procedures that are the subject of this clinical study. The study will feature two sequential arms with a companion registry of non-robotic participants to compare outcomes and quality of life between each robotic approach and standard of care. The procedures included in each arm are:

* Arm 1: Sleeve Gastrectomy, Cholecystectomy, Splenectomy, Hysterectomy, endometriosis, ureteral re-implant, and cervical and thoracic tracheoplasty, thymectomy, lobectomy/wedge lung resection, lung segmentectomy
* Arm 2: Bronchoplasty, Endoscopic Laryngeal/Pharyngeal Suturing, including: Vocal Feminization, Laryngeal Cleft Repair, Endolaryngeal Adjacent Tissue Transfer, Pharyngoplasty; Ileocolonic Resections; Laryngoplasty with or without Graft; Proctectomy with Ileal Pouch-Anal Anastomosis (IPAA)
* Registry: The registry will recruit patients undergoing the procedures performed in Arm 1 and 2 who will be treated with current standard of care techniques instead of robotic surgery.

Patient enrollment and assessments associated with procedures identified in Arm 1 will be completed prior to any procedures to be performed in Arm 2. The registry will prospectively enroll and evaluate patients undergoing non-surgical procedures at any time during the study period.

Participants will be evaluated from the first pre-operative assessment to 7 weeks post-operative.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 6 - 21 years of age (weighing at least 15 kilograms)
2. Subject clinically diagnosed with a medical condition for which one of the study procedures is appropriate therapy and selected as the treatment of choice by the guardian and surgeon.
3. Subject without previous treatment using a robotic surgery device
4. Subject or their guardian is willing and able to provide written informed consent
5. Subject or their guardian is willing and able to comply with the study protocol requirements

Exclusion Criteria:

1. Subject with uncorrected coagulopathy
2. Subject has clinical requirement for primary open operative procedure
3. Subject is ASA 4 or 5 status
4. Subject is contraindicated for general anesthesia or surgery
5. Subject is mentally handicapped or has a psychological disorder or severe systemic illness that would preclude compliance with study requirements or ability to provide informed consent
6. Subject is pregnant or suspected to be pregnant

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Performance | Intraoperative
  Performance defined as the conversion to an open approach required to complete the procedure
Number of Subjects With Device-related Serious Adverse Events | Intraoperative
  Safety is determined by measuring the number of subjects that experience device-related serious adverse events

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory (PedsQL) score | From enrollment to the end of treatment follow-up at 7 weeks post-operative
  Score of questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital Stanford, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided